CLINICAL TRIAL: NCT02956122
Title: A Two-Part, Multi-Center, Prospective, Phase 2/3 Clinical Study to Evaluate the Safety and Efficacy of GLASSIA as an Add-On Biopharmacotherapy to Conventional Steroid Treatment in Subjects With Acute Graft-Versus-Host Disease With Lower Gastrointestinal Involvement
Brief Title: A Phase 2/3 Study of GLASSIA for the Treatment of Acute GvHD
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The decision to discontinue the study was based on business reasons.
Sponsor: Baxalta now part of Shire (Industry)
Collaborators: Kamada, Ltd. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 471501
Record Dates: First submitted 2016-10-24; First posted 2016-11-07 (Estimated); Results first posted 2019-04-24 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2020-12

CONDITIONS: Graft Versus Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — alpha 1-Antitrypsin; Methylprednisolone; Albumins; Serum Albumin, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Study Part 1 - All Participants - GLASSIA (Experimental): Participants to receive GLASSIA (intravenously) and methylprednisolone or equivalent steroid (either IV or oral per investigator discretion)
  Interventions: Biological: GLASSIA; Drug: methylprednisolone or equivalent steroid
- Study Part 2 - GLASSIA (Experimental): Participants to receive GLASSIA (intravenously) and methylprednisolone or equivalent steroid (either IV or oral per investigator discretion)
  Interventions: Biological: GLASSIA; Drug: methylprednisolone or equivalent steroid
- Study Part 2 - Albumin (Control) (Placebo Comparator): Participants to receive control (intravenously) and methylprednisolone or equivalent steroid (either IV or oral per investigator discretion)
  Interventions: Drug: methylprednisolone or equivalent steroid; Biological: Albumin

INTERVENTIONS:
Biological: GLASSIA — GLASSIA [Alpha1-Proteinase Inhibitor (Human)]
  Other Names: as alpha-1 antitrypsin; A1PI; alpha-1 proteinase inhibitor
  Arms: Study Part 1 - All Participants - GLASSIA; Study Part 2 - GLASSIA
Drug: methylprednisolone or equivalent steroid — The conventional steroid treatment (methylprednisolone or equivalent steroid) will be supplied by the investigators per their institutional practice.
Biological: Albumin — The control vials contain human albumin 20% in 50 mL normal saline solution in glass vials (for non-United States (US) Countries), or Flexbumin 25% in 50 mL in normal saline solution in plastic IV bags (for US).
  Other Names: Human Albumin
  Arms: Study Part 2 - Albumin (Control)

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of GLASSIA as an add-on biopharmacotherapy to standard-of-care steroid treatment as the first-line treatment in participants with acute GvHD with lower GI involvement.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged ≥18 years at the time of screening
2. Recipient of an hematopoietic stem cell transplantation (HSCT)
3. The disease indication for which the participant required HSCT must be in remission
4. Newly diagnosed acute graft-versus-host disease (GvHD), including lower Gastrointestinal (GI) involvement (modified International Bone Marrow Transplant Registry [IBMTR] Severity Stage 1 to 4 [>500 mL diarrhea/day]), with or without other organ system involvement.
5. Willing to undergo or must have had a lower GI biopsy within 7 days of informed consent to confirm GI GvHD. Biopsy results are not needed to initiate treatment; however, if biopsy results are not consistent with aGvHD, treatment with GLASSIA will be discontinued.
6. Participants must be receiving systemic corticosteroids. Treatment with methylprednisolone/systemic steroids must have been initiated within 72 hours prior to the first dose of study treatment after enrollment
7. Evidence of myeloid engraftment (absolute neutrophil count ≥0.5 x 10^9/L)
8. Lower GI GvHD manifested by diarrhea must have other causes of diarrhea ruled out (eg, negative for Clostridium difficile or cytomegalovirus [CMV] infection or oral magnesium administration)
9. Karnofsky Performance Score ≥50%
10. If female of childbearing potential, participant presents with a negative blood pregnancy test
11. Females of childbearing potential with a fertile male sexual partner must agree to employ adequate contraception for the duration of the study.
12. Males must use adequate contraception and must not donate sperm for the duration of the study.
13. Participant is willing and able to comply with the requirements of the protocol

Exclusion Criteria:

1. Participant with manifestations of chronic GvHD
2. Participant with acute/chronic GvHD overlap syndrome
3. Participant whose GvHD developed after donor lymphocyte infusion
4. Participant with myocardial infarction within 6 months prior to enrollment or New York Heart Association Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to the first dose of study treatment, any electrocardiogram (ECG) abnormality at screening must be documented by the investigator as not medically relevant
5. Participant with evidence of recurrent malignancy
6. Participant with veno-occlusive disease (ie, sinusoidal obstruction syndrome)
7. Participant receiving GvHD treatment other than continued prophylaxis (eg, cyclosporine and/or mycophenolate mofetil, etc) or corticosteroid therapy. In addition, a participant who received the first dose of corticosteroid therapy for acute GvHD with lower GI involvement more than 72 hours before the first dose of study treatment is not eligible for the study
8. Participant with severe sepsis involving at least 1 organ failure
9. Participant who is seropositive or positive in the nucleic acid test for human immunodeficiency virus (HIV)
10. Participant with active hepatitis B or C
11. Participant has participated in another clinical study involving an investigational product (IP) or investigational device within 30 days prior to enrollment or is scheduled to participate in another clinical study involving an IP or investigational device during the course of this study
12. If female, participant is pregnant or lactating at the time of enrollment, or has plans to become pregnant during the study
13. Participant with a serious medical or psychiatric illness likely to interfere with participation in the study
14. Participant is a family member or employee of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2018-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (1):
- Georgia Cancer Center, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the low number of study participants).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted between 26 April 2017 (first participant first visit) and 03 May 2018 (last participant last visit).
Pre-assignment Details: A total of 1 participant was enrolled and completed Part 1 (GLASSIA) of the study, and was analyzed for efficacy and safety with individual PK parameters estimated. Part 2 (GLASSIA versus albumin [control]) was not initiated following discontinuation of the study due to operational and business considerations.
Groups:
- GLASSIA: Participants received an intravenous (IV) infusion of GLASSIA at a dose of 90 milligrams per kilogram (mg/kg) on Day 1 followed by 30 mg/kg every other day (Days 3 to 13), then followed by 120 mg/kg weekly (Days 15 to 50) along with 2 milligrams per kilogram per day (mg/kg/day) of methylprednisolone or equivalent steroid.
Period: Overall Study
Arm/Group | GLASSIA
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- GLASSIA: Participants received an IV infusion of GLASSIA at a dose of 90 mg/kg on Day 1 followed by 30 mg/kg every other day (Days 3 to 13), then followed by 120 mg/kg weekly (Days 15 to 50) along with 2 mg/kg/day of methylprednisolone or equivalent steroid.
Arm/Group | GLASSIA
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Overall Response (OR) At Day 28
Description: OR was defined as graft-versus-host disease (GvHD) complete response (CR) + partial response (PR), defined as: - GvHD CR was complete resolution of all signs and symptoms of acute GvHD in all organs without intervening salvage and GvHD PR was improvement of 1 stage in 1 or more organs involved in GvHD without progression in other organs.
Time Frame: Day 28
Population: Efficacy analysis set included all participants who were evaluated for overall response at Day 28. Participants who received at least 1 dose of study treatment and who had a lower GI biopsy that was consistent with acute GvHD were considered evaluable.
Measure: Number; unit: Percentage of participants
Arm/Group | GLASSIA
Number analyzed (Participants) | 1
Percentage of participants | 100

2. Secondary Outcome: Percentage of Participants Achieving Gastrointestinal (GI) Response at Day 28
Description: GI response was defined as complete response (CR) + partial response (PR), defined as: - GI CR was able to eat; not requiring parenteral nutrition, and passing primarily formed stools - GI PR was decrease in need for parenteral nutrition to less than or equal to (<=) 50% of required calories; and reduction of stool volume by greater than or equal to (>=) 50%, without ileus.
Time Frame: Day 28
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | GLASSIA
Number analyzed (Participants) | 1
Percentage of participants | 100

3. Secondary Outcome: Percentage of Participants Achieving Overall Response at Day 56
Description: Overall response was defined as graft-versus-host disease (GvHD) complete response (CR) + partial response (PR), defined as: - GvHD CR was complete resolution of all signs and symptoms of acute GvHD in all organs without intervening salvage - GvHD PR was improvement of 1 stage in 1 or more organs involved in GvHD without progression in other organs.
Time Frame: Day 56
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | GLASSIA
Number analyzed (Participants) | 1
Percentage of participants | 100

4. Secondary Outcome: Acute Graft-versus-host Disease (GvHD) Grading at Days 28, 56 and 180
Description: Grading of GvHD was performed by the investigator according to the modified International Bone Marrow Transplant Registry (IBMTR) grading system which classifies the degree of involvement of each organ system by stage on a scale of 0 to 4. The degree of skin involvement was staged depending upon degree and severity of the lesions: Stage 1: Maculopapular rash over less than (<) 25% of body area, Stage 2: Maculopapular rash over 25 to 50% of body area, Stage 3: Generalized erythroderma, Stage 4: Generalized erythroderma with bullous formation. Degree of GI involvement was staged based on severity of diarrhoea: Stage 1: 500 to 1000 mL/day,Stage 2: 1000 to 1500 mL/day, Stage 3: 1500 to 2000 mL/day, Stage 4: greater than (>) 2000 mL/day OR pain OR ileus. Degree of liver involvement was staged based upon serum total bilirubin level as follows: Stage 1: 2 to 3 mg/dL, Stage 2: 3 to 6 mg/dL, Stage 3: 6 to 15 mg/dL, Stage 4: >15 mg/dL.
Time Frame: Days 28, 56 and 180
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GLASSIA
Number analyzed (Participants) | 1
Participants
  Day 28: Degree of skin Involvement: Stage 0 | 1
  Day 28: Degree of skin Involvement: Stage 1 | 0
  Day 28: Degree of skin Involvement: Stage 2 | 0
  Day 28: Degree of skin Involvement: Stage 3 | 0
  Day 28: Degree of skin Involvement: Stage 4 | 0
  Day 28: Degree of GI Involvement: Stage 0 | 1
  Day 28: Degree of GI Involvement: Stage 1 | 0
  Day 28: Degree of GI Involvement: Stage 2 | 0
  Day 28: Degree of GI Involvement: Stage 3 | 0
  Day 28: Degree of GI Involvement: Stage 4 | 0
  Day 28: Degree of liver Involvement: Stage 0 | 1
  Day 28: Degree of liver Involvement: Stage 1 | 0
  Day 28: Degree of liver Involvement: Stage 2 | 0
  Day 28: Degree of liver Involvement: Stage 3 | 0
  Day 28: Degree of liver Involvement: Stage 4 | 0
  Day 56: Degree of skin Involvement: Stage 0 | 1
  Day 56: Degree of skin Involvement: Stage 1 | 0
  Day 56: Degree of skin Involvement: Stage 2 | 0
  Day 56: Degree of skin Involvement: Stage 3 | 0
  Day 56: Degree of skin Involvement: Stage 4 | 0
  Day 56: Degree of GI Involvement: Stage 0 | 1
  Day 56: Degree of GI Involvement: Stage 1 | 0
  Day 56: Degree of GI Involvement: Stage 2 | 0
  Day 56: Degree of GI Involvement: Stage 3 | 0
  Day 56: Degree of GI Involvement: Stage 4 | 0
  Day 56: Degree of liver Involvement: Stage 0 | 1
  Day 56: Degree of liver Involvement: Stage 1 | 0
  Day 56: Degree of liver Involvement: Stage 2 | 0
  Day 56: Degree of liver Involvement: Stage 3 | 0
  Day 56: Degree of liver Involvement: Stage 4 | 0
  Day 180: Degree of skin Involvement: Stage 0 | 1
  Day 180: Degree of skin Involvement: Stage 1 | 0
  Day 180: Degree of skin Involvement: Stage 2 | 0
  Day 180: Degree of skin Involvement: Stage 3 | 0
  Day 180: Degree of skin Involvement: Stage 4 | 0
  Day 180: Degree of GI Involvement: Stage 0 | 1
  Day 180: Degree of GI Involvement: Stage 1 | 0
  Day 180: Degree of GI Involvement: Stage 2 | 0
  Day 180: Degree of GI Involvement: Stage 3 | 0
  Day 180: Degree of GI Involvement: Stage 4 | 0
  Day 180: Degree of liver Involvement: Stage 0 | 1
  Day 180: Degree of liver Involvement: Stage 1 | 0
  Day 180: Degree of liver Involvement: Stage 2 | 0
  Day 180: Degree of liver Involvement: Stage 3 | 0
  Day 180: Degree of liver Involvement: Stage 4 | 0

5. Secondary Outcome: Incidence of Chronic Graft-versus-host Disease (GvHD)
Description: Incidence of chronic GvHD at Days 180 and 365 was reported.
Time Frame: Days 180 and 365
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | GLASSIA
Number analyzed (Participants) | 1
Participants
  Day 180 | 0
  Day 365 | 0

6. Secondary Outcome: Duration of Overall Response (OR)
Description: OR was defined as GvHD CR + PR, defined as: - GvHD CR was complete resolution of all signs and symptoms of acute GvHD in all organs without intervening salvage - GvHD PR was improvement of 1 stage in 1 or more organs involved in GvHD without progression in other organs. Duration of OR was not assessed due to the termination of the study.
Time Frame: Baseline up to Day 365
Population: Efficacy analysis set included all participants who were evaluated for overall response at Day 28. Participants who received at least 1 dose of study treatment and who had a lower GI biopsy that was consistent with acute GvHD were considered evaluable. Here, number of participants analyzed refer to the participants evaluable for this outcome.
Arm/Group | GLASSIA
Number analyzed (Participants) | 0

7. Secondary Outcome: Duration of Gastrointestinal (GI) Response
Description: GI response was defined as CR + PR, defined as: - GI CR was able to eat; not requiring parenteral nutrition, and passing primarily formed stools - GI PR was decrease in need for parenteral nutrition to <= 50% of required calories; and reduction of stool volume by >= 50%, without ileus. Duration of GI response was not assessed due to the termination of the study.
Time Frame: Baseline up to Day 365
Population: as for outcome 6
Arm/Group | GLASSIA
Number analyzed (Participants) | 0

8. Secondary Outcome: Overall Survival (OS) - Percentage of Participants With an Event
Description: OS was defined as the time from the date of randomization to the date of death due to any cause.
Time Frame: Days 100, 180 and 365
Population: Safety analysis (SAF) set consisted of all participants who received at least 1 dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | GLASSIA
Number analyzed (Participants) | 1
Percentage of participants
  Day 100 | NA — No deaths were observed during the study.
  Day 180 | NA — No deaths were observed during the study.
  Day 365 | NA — No deaths were observed during the study.

9. Secondary Outcome: Transplant-related Mortality
Description: Transplant-related mortality was determined by the investigator (any deaths considered related to the transplant).
Time Frame: Days 28, 56, 100 and 180
Population: SAF set consisted of all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | GLASSIA
Number analyzed (Participants) | 1
Participants
  Day 28 | 0
  Day 56 | 0
  Day 100 | 0
  Day 180 | 0

10. Secondary Outcome: Failure-free Survival - Percentage of Participants With an Event
Description: Failure-free survival was defined as the absence of all of the following criteria: Need for second-line treatment for acute GvHD, Non-relapse mortality (death during continuous complete remission) and recurrent malignancy.
Time Frame: Days 100 and 180
Population: SAF set consisted of all participants who received at least 1 dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | GLASSIA
Number analyzed (Participants) | 1
Percentage of participants
  Day 100 | 100
  Day 180 | 100

11. Secondary Outcome: Graft-versus-host Disease (GvHD)-Free Survival - Percentage of Participants With an Event
Description: GVHD-free survival was defined as being alive without previous onset of acute GVHD or chronic GVHD requiring immunosuppressive therapy.
Time Frame: Days 28, 56, 100, 180 and 365
Population: SAF set consisted of all participants who received at least 1 dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | GLASSIA
Number analyzed (Participants) | 1
Percentage of participants
  Day 28 | 100
  Day 56 | 100
  Day 100 | 100
  Day 180 | 100
  Day 365 | 100

12. Secondary Outcome: Infection-related Mortality - Percentage of Participants With an Event
Description: Infection-related mortality was determined by the investigator (any deaths considered related to infection [including infections related to hematopoietic stem cell transplant {HSCT}]).
Time Frame: Days 28, 56, 100 and 180
Population: SAF set consisted of all participants who received at least 1 dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | GLASSIA
Number analyzed (Participants) | 1
Percentage of participants
  Day 28 | 0
  Day 56 | 0
  Day 100 | 0
  Day180 | 0

13. Secondary Outcome: Graft-versus-host Disease (GvHD)-Related Mortality - Percentage of Participants With an Event
Description: Graft-versus-host disease (GvHD)-related mortality was determined by the investigator (any deaths considered related to GvHD).
Time Frame: Days 28, 56, 100 and 180
Population: SAF set consisted of all participants who received at least 1 dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | GLASSIA
Number analyzed (Participants) | 1
Percentage of participants
  Day 28 | 0
  Day 56 | 0
  Day 100 | 0
  Day 180 | 0

14. Secondary Outcome: All-cause Mortality - Percentage of Participants With an Event
Description: All-cause mortality was defined as the time from HSCT to death due to any cause.
Time Frame: Days 28, 56, 100 and 180
Population: SAF set consisted of all participants who received at least 1 dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | GLASSIA
Number analyzed (Participants) | 1
Percentage of participants
  Day 28 | 0
  Day 56 | 0
  Day 100 | 0
  Day180 | 0

15. Secondary Outcome: Number of Participants With Adverse Events (AEs), Treatment-related AEs, Serious Adverse Events (SAEs), Treatment-related SAEs and Temporally-associated AEs
Description: An AE was defined as any untoward medical occurrence in a participant administered an investigational product (IP) that does not necessarily have a causal relationship with the treatment. An SAE was defined as an untoward medical occurrence that at any dose meets one or more of the following criteria: outcome was fatal/results in death, life-threatening, required inpatient hospitalization or resulted in prolongation of an existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event.
Time Frame: From start of study drug administration up to 371 days
Population: SAF set consisted of all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | GLASSIA
Number analyzed (Participants) | 1
Participants
  Any Adverse Event | 1
  Treatment-related AEs | 0
  Serious adverse Events (SAEs) | 0
  Treatment-related SAEs | 0
  Temporally-associated AEs | 0

16. Secondary Outcome: Number of Participants With Clinically Significant Changes in Clinical Laboratory Assessments
Description: Clinical laboratory assessments such as hematology, clinical chemistry, lipid and coagulation panels and urinalysis were performed.
Time Frame: Baseline up to Day 56
Population: SAF set consisted of all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | GLASSIA
Number analyzed (Participants) | 1
Participants | 0

17. Secondary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs
Description: Vital signs included body temperature, respiratory rate, pulse rate and systolic and diastolic blood pressure.
Time Frame: Baseline up to Day 56
Population: SAF set consisted of all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | GLASSIA
Number analyzed (Participants) | 1
Participants | 0

18. Secondary Outcome: Number of Participants With Recurrence of Primary Malignancies
Description: Incidence of recurrence of primary malignancies was reported.
Time Frame: Baseline up to Day 365
Population: SAF set consisted of all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | GLASSIA
Number analyzed (Participants) | 1
Participants | 0

19. Secondary Outcome: Area Under the Plasma Concentration Curve (AUC0-inf) From Time Zero to Infinity
Description: AUC of GLASSIA was reported.
Time Frame: Day 1: through 48 hours; Day 13: through 48 hours; Day 22 and Day 50: through approximately 168 hours
Population: PK Analysis set included all participants in the SAF set who have at least 1 PK or stool sample collected.
Measure: Number; unit: Hour*milligrams per deciliter (h*mg/dL)
Groups:
- GLASSIA: Day 1: 90 mg/kg: Participants received an IV infusion of 90 mg/kg GLASSIA.
- GLASSIA: Day 13: 30 mg/kg: Participants received an IV infusion of 30 mg/kg GLASSIA.
- GLASSIA: Day 22: 120 mg/kg; GLASSIA: Day 50: 120 mg/kg: Participants received an IV infusion of 120 mg/kg GLASSIA.
Arm/Group | GLASSIA: Day 1: 90 mg/kg | GLASSIA: Day 13: 30 mg/kg | GLASSIA: Day 22: 120 mg/kg | GLASSIA: Day 50: 120 mg/kg
Number analyzed (Participants) | 1 | 1 | 1 | 1
Hour*milligrams per deciliter (h*mg/dL) | 61500 | 43500 | 126000 | 117000

20. Secondary Outcome: Area Under the Plasma Concentration Curve From Time Zero to Time "t" AUC(0-t) of GLASSIA
Description: AUC(0-t) of GLASSIA was reported.
Time Frame: Day 1: through 48 hours, Day 13: through 48 hours, Day 22 and Day 50: through approximately 168 hours
Population: PK Analysis set included all participants in the SAF set who have at least 1 PK or stool sample collected.
Measure: Number; unit: h*mg/dL
Arm/Group | GLASSIA: Day 1: 90 mg/kg | GLASSIA: Day 13: 30 mg/kg | GLASSIA: Day 22: 120 mg/kg | GLASSIA: Day 50: 120 mg/kg
Number analyzed (Participants) | 1 | 1 | 1 | 1
h*mg/dL | 16300 | 11000 | 40400 | 33400

21. Secondary Outcome: Systemic Clearance at Steady State (CLss) of GLASSIA
Description: CLss of GLASSIA was reported.
Time Frame: Day 1: through 48 hours, Day 13: through 48 hours, Day 22 and Day 50: through approximately 168 hours
Population: PK Analysis set included all participants in the SAF set who have at least 1 PK or stool sample collected.
Measure: Number; unit: Deciliters per hour (dL/h)
Arm/Group | GLASSIA: Day 13: 30 mg/kg | GLASSIA: Day 22: 120 mg/kg | GLASSIA: Day 50: 120 mg/kg
Number analyzed (Participants) | 1 | 1 | 1
Deciliters per hour (dL/h) | 0.297 | 0.286 | 0.260

22. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of GLASSIA
Description: Cmax of GLASSIA was reported.
Time Frame: Day 1: through 48 hours, Day 13: through 48 hours, Day 22 and Day 50: through approximately 168 hours
Population: PK Analysis set included all participants in the SAF set who have at least 1 PK or stool sample collected.
Measure: Number; unit: Milligrams per deciliter (mg/dl)
Arm/Group | GLASSIA: Day 1: 90 mg/kg | GLASSIA: Day 13: 30 mg/kg | GLASSIA: Day 22: 120 mg/kg | GLASSIA: Day 50: 120 mg/kg
Number analyzed (Participants) | 1 | 1 | 1 | 1
Milligrams per deciliter (mg/dl) | 339 | 262 | 390 | 409

23. Secondary Outcome: Apparent Volume of Distribution at Steady State (Vss) of GLASSIA
Description: Vss of GLASSIA was reported.
Time Frame: Day 1: through 48 hours, Day 13: through 48 hours, Day 22 and Day 50: through approximately 168 hours
Population: PK Analysis set included all participants in the SAF set who have at least 1 PK or stool sample collected.
Measure: Number; unit: Deciliter (dL)
Arm/Group | GLASSIA: Day 13: 30 mg/kg | GLASSIA: Day 22: 120 mg/kg | GLASSIA: Day 50: 120 mg/kg
Number analyzed (Participants) | 1 | 1 | 1
Deciliter (dL) | 50.9 | 123 | 91.1

24. Secondary Outcome: Apparent Terminal Half-life (t1/2) of GLASSIA
Description: Apparent terminal half-life (hour), determined as ln2/lambda-z. lambda-z is the apparent terminal rate constant (one per hour), determined by linear regression of the terminal points of the log-linear concentration-time curve. Visual assessment will be used to identify the terminal linear phase of the concentration-time profile. A minimum of 3 data points will be used for determination. t1/2 of GLASSIA was reported.
Time Frame: Day 1: through 48 hours, Day 13: through 48 hours, Day 22 and Day 50: through approximately 168 hours
Population: PK Analysis set included all participants in the SAF set who have at least 1 PK or stool sample collected.
Measure: Number; unit: Hour (h)
Arm/Group | GLASSIA: Day 1: 90 mg/kg | GLASSIA: Day 13: 30 mg/kg | GLASSIA: Day 22: 120 mg/kg | GLASSIA: Day 50: 120 mg/kg
Number analyzed (Participants) | 1 | 1 | 1 | 1
Hour (h) | 152 | 117 | 317 | 247

25. Secondary Outcome: Mean Residence Time (MRT) of GLASSIA
Description: MRT of GLASSIA was not calculated.
Time Frame: Day 1: through 48 hours, Day 13: through 48 hours, Day 22 and Day 50: through approximately 168 hours
Population: PK Analysis set included all participants in the SAF set who have at least 1 PK or stool sample collected. Her, the number of participants analyzed refer to the participants evaluable for this outcome at specified time point.
Arm/Group | GLASSIA: Day 1: 90 mg/kg | GLASSIA: Day 13: 30 mg/kg | GLASSIA: Day 22: 120 mg/kg | GLASSIA: Day 50: 120 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0

26. Secondary Outcome: Trough Plasma Concentration at Steady State (Ctrough) of GLASSIA
Description: Ctrough of GLASSIA was not assessed due to the termination of the study.
Time Frame: Day 1: through 48 hours, Day 13: through 48 hours, Day 22 and Day 50: through approximately 168 hours
Population: PK Analysis set included all participants in the SAF set who have at least 1 PK or stool sample collected. Here, number of participants analyzed refer to the participants evaluable for this outcome at specified time point.
Arm/Group | GLASSIA: Day 1: 90 mg/kg | GLASSIA: Day 13: 30 mg/kg | GLASSIA: Day 22: 120 mg/kg | GLASSIA: Day 50: 120 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the start of drug administration up to 371 days
Arm/Group | GLASSIA
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLASSIA (N=1)
Platelet count decreased/ (Investigations) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (6)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2)
Weight decreased (Investigations) | 1 (1)
Blood cholesterol increased (Investigations) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Hot flush (Vascular disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
White blood cell count decreased (Investigations) | 1 (3)
Injection site reaction (General disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (2)
Mucosal infection (Infections and infestations) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Localised oedema (General disorders) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (2)
Cellulitis (Infections and infestations) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Bilirubin conjugated increased (Investigations) | 1 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Neutrophil count decreased (Investigations) | 1 (1)
Tongue ulceration (Gastrointestinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonmentor termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2017-04-19): https://cdn.clinicaltrials.gov/large-docs/22/NCT02956122/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-13): https://cdn.clinicaltrials.gov/large-docs/22/NCT02956122/SAP_001.pdf